CLINICAL TRIAL: NCT04207450
Title: Effect of Glutaraldehyde on Dentin Hypersensitivity After Non-surgical Periodontal Treatment: a Triple-blind Randomized Clinical Trial.
Brief Title: Effect of Glutaraldehyde on Dentin Hypersensitivity After Non-surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Clinical Professor, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFPara-006
Record Dates: First submitted 2019-12-16; First posted 2019-12-20 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Dentin Sensitivity
Keywords: Clinical trials; Dentin Sensitivity; glutaraldehyde; Desensitizing agents
MeSH Terms: conditions — Dentin Sensitivity | interventions — phosphoric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo Group (Placebo Comparator): Placebo Gel + Placebo Solution (Distilled Water)
  Interventions: Other: Placebo gel
- Placebo Gel + Glutaraldehyde (GPG) (Experimental): Placebo Gel + 5% Glutaraldehyde Aqueous Solution
  Interventions: Other: Placebo Gel + 5% Glutaraldehyde Aqueous Solution
- Phosphoric Acid + Glutaraldehyde (GAG) (Experimental): 37% Phosphoric Acid + Glutaraldehyde Aqueous Solution (GAG)
  Interventions: Other: Phosphoric Acid 37% + Solução aquosa de glutaraldeído a 5%

INTERVENTIONS:
Other: Placebo gel — Placebo gel application followed by placebo solution application (distilled water)
  Arms: Placebo Group
Other: Placebo Gel + 5% Glutaraldehyde Aqueous Solution — Placebo gel followed by 5% aqueous glutaraldehyde solution
  Arms: Placebo Gel + Glutaraldehyde (GPG)
Other: Phosphoric Acid 37% + Solução aquosa de glutaraldeído a 5% — 37% phosphoric acid application followed by 5% aqueous glutaraldehyde solution
  Arms: Phosphoric Acid + Glutaraldehyde (GAG)

SUMMARY:
This randomized, placebo-controlled, triple-blind trial aims to evaluate the effect of glutaraldehyde associated or not with 37% phosphoric acid conditioning on dentin hypersensitivity reduction after non-surgical periodontal treatment, and its durability after 15 and 30 days. desensitizing treatment. Additionally, investigate the impact of these treatments on health-related quality of life. The investigators selected patients who, after scraping and planing procedures, presented at least 2 teeth meeting the following inclusion criteria: presence of gingival recession without or with a periodontal pocket up to 5mm probing depth, which presented painful sensitivity response to tactile stimulus. and evaporative. Subjects were randomized into 3 groups: Placebo Group (GP) - Placebo Gel application followed by Placebo solution (distilled water); GPG- Placebo Gel application followed by application 5% aqueous glutaraldehyde solution; GSG - Application of 37% phosphoric acid followed by 5% aqueous glutaraldehyde solution. The sensitivity of the dental elements was evaluated by pain stimuli (tactile and evaporative) with the aid of a Visual Analog Scale (VAS). A questionnaire was applied to patients with the objective of capturing psychosocial experiences, prior to treatment and one month after its completion, to assess the impact of desensitizing treatment on health-related quality of life. Data will be collected and appropriate statistical tests will be applied.

ELIGIBILITY:
Inclusion Criteria:

- Presence of gingival recession without or with periodontal pocket up to 5mm probing depth, which presented painful sensitivity response to tactile and evaporative stimuli.

Exclusion Criteria:

* Systemic diseases;
* Pulpitis;
* Carious lesions;
* Presence of restorations in selected teeth;
* Cracked enamel;
* Noncarious cervical lesions;
* Use of medication with analgesics and/or anti-inflammatories;
* Pregnant or lactating women;
* Desensitizing treatment and periodontal treatment received during three months prior to study recruitment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Dentin sensitivity | Immediately after the intervention
  Evaluation of pain (dentin sensitivity) by applying tactile (exploratory probe pressure) and evaporative (air blast) stimuli on exposed dentin. Sensitivity will be measured using the Thomas Schiff scale from 0 to 3. Zero means absent dentin sensitivity and three means severe dentin sensitivity.

SECONDARY OUTCOMES:
Dentin hypersensitivity experience questionnaire | Immediately after the intervention
  A self-reported questionnaire was applied by the patients with the objective of capturing psychosocial experiences, previous treatment and one month after its completion, aiming to evaluate the impact of desensitizing treatment on health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Para, Belém, Pará, Brazil